CLINICAL TRIAL: NCT00727259
Title: Evaluation of Satisfaction in Patients Receiving PegIntron Pen/Rebetol for Hepatitis C
Brief Title: Evaluation of Satisfaction in Patients Receiving PegIntron Pen/Rebetol for Hepatitis C (Study P04067)
Acronym: SATISFACTION
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04067
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2009-08-06 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with chronic hepatitis C: Adult patients with chronic hepatitis C treated with PegIntron pen/Rebetol.
  Interventions: Biological: Peginterferon alfa-2b (SCH 54031); Drug: Ribavirin (SCH 18908)

INTERVENTIONS:
Biological: Peginterferon alfa-2b (SCH 54031) — Peginterferon alfa-2b will be administered according to the products' labeling.
  Other Names: PegIntron; PegPen
Drug: Ribavirin (SCH 18908) — Ribavirin will be administered according to the products' labeling.
  Other Names: Rebetol

SUMMARY:
The current gold standard for treatment of chronic hepatitis C (CHC) patients is with pegylated interferon plus ribavirin. Drug administration accuracy and ease of use will definitely determine treatment effectiveness. This is the idea behind the development and usage of the PegPen. The goal of this study is to determine the satisfaction grade with this novel device.

DETAILED DESCRIPTION:
Enrollment of patients will occur in a sequential order of treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with hepatitis C

Exclusion Criteria:

* According to the products' labeling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic hepatitis C treated with PegIntron pen/Rebetol at sites in France.
Sampling Method: Probability Sample
Enrollment: 1995 (Actual)
Dates: Start 2004-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled: 1995 subjects; all questionnaires were returned for 940 subjects.
Period: Overall Study
Arm/Group | Patients With Chronic Hepatitis C
Started | 1995
Completed | 940
Not Completed | 1055
Not completed — Not all questionnaires completed | 1055

BASELINE CHARACTERISTICS:
Groups:
- Patients With Chronic Hepatitis C: Adult patients with chronic hepatitis C treated with PegIntron pen/Rebetol. Results presented concern only participants with all questionnaires returned (940).
Arm/Group | Patients With Chronic Hepatitis C
Number analyzed (Participants) | 940
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.50 (12.34)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 323
  Male | 616
  Missing data | 1
Region of Enrollment [Number; unit: Participants]
  France | 940

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Satisfaction of the PegPen (PegIntron Preparation and Injection Easiness) Using a Patient Questionnaire Answered at 1 Month and 3 Months
Description: Patient satisfaction for each item on the questionnaires was rated on a scale from 0 (not satisfied) to 7 (very satisfied).
Time Frame: The patient was instructed to answer and return by mail the first self-questionnaire after 1 month of treatment and the second one after 3 months of treatment.
Population: Both patient questionnaires were returned by 940 subjects. However, some items were not rated on the returned questionnaires. The missing data for questionnaire items range from 24 subjects to 72 subjects.
Measure: Mean (Standard Deviation); unit: satisfaction rating from 0-7
Groups:
- After 1 Month of Treatment; After 3 Months of Treatment: Adult patients with chronic hepatitis C treated with PegIntron pen/Rebetol.
Arm/Group | After 1 Month of Treatment | After 3 Months of Treatment
Number analyzed (Participants) | 940 | 940
satisfaction rating from 0-7
  Ease of preparation of the Pen | 5.48 (1.74) | 5.91 (1.41)
  Simplicity of adjustment of the injected dose | 5.74 (1.71) | 6.08 (1.41)
  Time required for the preparation of the injection | 5.49 (1.52) | 5.84 (1.32)
  Ease of injection | 5.89 (1.46) | 6.00 (1.37)
  Characteristics of the needle | 6.14 (1.25) | 6.25 (1.21)
  Overall satisfaction with the system of injection | 5.99 (1.73) | 6.04 (1.32)

ADVERSE EVENTS:
Description: Per protocol, non-serious adverse events and serious adverse events were not required to be captured as part of the study database, therefore, none were collected, and the number at risk is zero.
Arm/Group | Patients With Chronic Hepatitis C
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or communication (written or oral) could be performed by the Principal Investigator only after written approval from Schering-Plough.